CLINICAL TRIAL: NCT02888457
Title: Assessment of the Nasopharyngeal Carriage of Streptococcus Pneumoniae (Sp) and Other Common Pathogens in Infants (6-30 Months of Age) With Acute Otitis Media and in Healthy Infants (6-30 Months of Age) Attending Day-care Centers
Brief Title: Carriage of Streptococcus Pneumoniae in Infants With Acute Otitis Media and in Infants Attending Day-care Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Van Damme (Other)
Collaborators: Centre Hospitalier Intercommunal Creteil (Other); University of Bristol (Other); University Ghent (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Sponsor-Investigator, Pierre Van Damme, Prof, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15/45/471
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Streptococcus Pneumoniae; Nasopharyngeal Carriage
Keywords: nasopharyngeal carriage; Streptococcus pneumoniae; acute otitis media; day-care centers
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AOM (acute otitis media) (Other): Infants (6-30 months of age) with acute otitis media
  Interventions: Other: Nasopharyngeal sampling with a swab
- DCC (day-care centers) (Other): Healthy infants (6-30 months of age) attending day-care centers
  Interventions: Other: Nasopharyngeal sampling with a swab

INTERVENTIONS:
Other: Nasopharyngeal sampling with a swab

SUMMARY:
Rationale

In Belgium, a unique situation exists for two reasons: on the one hand, the pneumococcal conjugate vaccine (PCV) program, which started in 2007, has quickly reached high coverage in infants: 3-dose coverage rose from 89 % in 2008 to 96.5 % in 2012 in Flanders and from 80.7 % in 2009 to 89.2 % in 2012 in Wallonia; and on the other hand, serotype coverage has moved from PCV7 (since 2007) to PCV13 (since 2011) and very recently to PCV10 (since July 2015 in Flanders and expected in May 2016 in the French Community). Invasive pneumococcal disease (IPD) surveillance has demonstrated a major impact on PCV13 serotypes in infants < 2 years of age. The impact of the current change in PCV-program is hard to predict, but could eventually result in a re-emergence of serotypes not covered by PCV10 (i.e. 3, 6A and 19A).

With this unique situation the foundation was laid for a carriage study during which the nasopharyngeal carriage of Streptococcus pneumonia (Sp) and other common colonizers of the nasopharynx will be studied in infants with acute otitis media (AOM) and in healthy infants attending day-care centers (DCC), two populations with high reported pneumococcal carriage. Young children are an important reservoir and major source of transmission of bacteria to the whole community and thus the preferred population to study nasopharyngeal (NP) carriage.

Aim of the study

The main aim of this study is to evaluate if changes in the conjugate anti-pneumococcal vaccination program in Belgium have an impact on the nasopharyngeal carriage of Pneumococcus in infants aged 6-30 months suffering from AOM or attending day-care, in order to guide future pneumococcal vaccine program decisions and vaccine development, and to feed AOM treatment guidelines in a PCV-program environment. The study will monitor overall pneumococcal carriage, the serotypes involved and the sensitivity of the isolated strains to antibiotics. In addition, the rhinopharyngeal carriage of other common nasopharyngeal colonizers associated with disease, in particular Haemophilus influenzae, will be studied in order to evaluate if changes in pneumococcal carriage impact on the carriage of those pathogens. In infants with AOM, the study will also monitor the clinical course of the AOM and a second nasopharyngeal sample will be taken in case of antibiotic treatment failure or AOM recurrence to identify any association with the carried pathogen.

DETAILED DESCRIPTION:
Study populations

Two infant populations with high (50 % and more) reported carriage of Sp were identified and will be approached for this study:

1. Infants aged 6-30 months presenting with acute otitis media (according to specific clinical and otoscopic criteria) at their first line general physician or paediatrician and who have not recently received antibiotics and have no severe underlying disease (AOM infants).
2. Healthy infants aged 6-30 months attending a day-care center and not recently having received antibiotics (DCC infants).

Investigator(s), study sites

75-87 paediatricians and general practitioners (GPs), and approximately 75 DCC throughout the whole of Belgium. Paediatricians in first line hospitals are allowed to participate.

The Primary objective

is to detect significant prevalence change of Sp serotypes 19A or 6A carriage over the observation period (three years, 2016-2018) in each of both study populations (AOM or DCC infants).

Number of subjects

In the first year (2016), 700 and from the second year ( 2016-2017) onward 900, patients with AOM (between the ages of 6 and 30 months) will be included every year. The same number of healthy infants attending DCC will be included each year. Sample size was calculated to allow comparison between children recruited in the first winter season, who have received PCV13 for all or the majority of their pneumococcal vaccinations, and the children in the following seasons, who will have received PCV10 for the majority or all of their pneumococcal vaccinations. Some over-recruitment will be done during the first winter (2016) of infants vaccinated in the region that has not yet changed from PCV13 to PCV10, since these infants will have received PCV13 for their 12 months booster too. The proposed sample size allows to detect changes as low as 3 % for 19A and 6A combined, and 4 % for each of them separately with 80 % power, in each of the AOM and day-care infant groups.

Period of observation

Since Sp carriage as well as AOM are most prevalent in and around the winter season, recruitment will be scheduled focusing on this period. In 2016, recruitment of infants presenting with AOM is foreseen from January till end of May, but can be extended to June if necessary to achieve the target number. Thereafter, infants with AOM will be recruited every year from October till end of May (starting October 2016). For healthy infants attending DCC recruitment is planned to start in March 2016, and thereafter every season from October 1st till May 31st. The current protocol covers the first observation period, from 2016 to 2018 covering 3 winter seasons.

ELIGIBILITY:
Inclusion Criteria AOM:

* Informed consent read and signed AND acute onset of AOM symptoms within the preceding 7 days AND otoscopic signs OR new onset otorrhea not due to otitis externa

Inclusion Criteria DCC:

* Informed consent read and signed AND residing in a day-care center with a minimum of 9 infants daily present

Exclusion Criteria:

* Having received antibiotics in the past 7 days AND/OR a severe associated pathology AND/OR infant already included in the same winter season AND/OR (for infants recruited in hospital) referral by GP or having received 3 or more antibiotic treatments in the past 3 months

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2817 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
prevalence | 3 years
  To detect significant prevalence change of Sp serotypes 19A or 6A carriage over the observation period (three years, 2016-2018) in each of both study populations (AOM or DCC infants).

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Theeten, Professor, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van den Bosch E, Vermeulen H, Ekinci E, Paranthoen L, Van Heirstraeten L, Malhotra-Kumar S, Desmet S, Theeten H, Maertens K. Interplay between maternal Tdap and infant pneumococcal vaccination in shaping infant pneumococcal vaccine serotype carriage. J Infect Dis. 2025 Aug 30:jiaf458. doi: 10.1093/infdis/jiaf458. Online ahead of print. PMID 40884828